CLINICAL TRIAL: NCT04944147
Title: Neuromodulation Through Brain Stimulation-assisted Cognitive Training in Patients With Post-COVID-19 Cognitive Impairment
Brief Title: Cognitive Training and Brain Stimulation in Patients With Post-COVID-19 Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Neuromod-COV
Record Dates: First submitted 2021-06-28; First posted 2021-06-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: COVID-19; Post-COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Transcranial Direct Current Stimulation; Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal tDCS + cognitive training (Experimental): device: anodal transcranial direct current stimulation (tDCS), 9 sessions with 20 minutes stimulation each (2 mA) over left dorsolateral prefrontal cortex
  behavioral: intensive cognitive training intensive cognitive training of letter memory updating task (20 minutes), 9 sessions
  Interventions: Device: Anodal tDCS; Behavioral: Intensive cognitive training
- Sham tDCS + cognitive training (Placebo Comparator): device: sham transcranial direct current stimulation (tDCS), 9 sessions with 30 seconds stimulation each (2 mA) over left dorsolateral prefrontal cortex
  behavioral: intensive cognitive training intensive cognitive training of letter memory updating task (20 minutes), 9 sessions
  Interventions: Device: Sham tDCS; Behavioral: Intensive cognitive training
- Sham tDCS + Progressive Muscle Relaxation training (Active Comparator): device: sham transcranial direct current stimulation (tDCS), 9 sessions with 30 seconds stimulation each (2 mA) over left dorsolateral prefrontal cortex
  behavioral: progressive muscle relaxation (PMR) standardized instructed PMR (20 minutes), 9 sessions
  Interventions: Device: Sham tDCS; Behavioral: Progressive muscle relaxation (PMR)

INTERVENTIONS:
Device: Anodal tDCS — Anodal transcranial direct current stimulation (tDCS), 9 sessions with 20 minutes stimulation each (2 mA)
  Arms: Anodal tDCS + cognitive training
Device: Sham tDCS — Sham transcranial direct current stimulation (tDCS), 9 sessions with 30 sec stimulation each (2 mA) to ensure blinding of participants
  Arms: Sham tDCS + Progressive Muscle Relaxation training; Sham tDCS + cognitive training
Behavioral: Intensive cognitive training — Intensive cognitive training of a letter memory updating task, 9 sessions
  Arms: Anodal tDCS + cognitive training; Sham tDCS + cognitive training
Behavioral: Progressive muscle relaxation (PMR) — Standardized instructed PMR training, 9 sessions
  Arms: Sham tDCS + Progressive Muscle Relaxation training

SUMMARY:
The aim of the study is to investigate effects of brain stimulation-assisted cognitive training in patients with persistent subjective or objective cognitive impairment after polymerase chain reaction (PCR)-positive COVID-19 disease.

DETAILED DESCRIPTION:
Long-term persistent symptoms occur in a substantial number of patients diagnosed with coronavirus 2019 disease (COVID-19). First evidence suggests that long-term symptoms develop not only after severe courses of the disease, but also after less serious illness and include various symptoms such as fatigue and impaired memory, concentration or sleep. During recovery, these symptoms present a heavy burden for patients, who then often experience psychological distress and reduced quality of life. The goal of the present study is to assess the effects of cognitive training alone or in combination with tDCS on cognitive performance, quality of life and mental health in patients with subjective or objective cognitive impairments following post-COVID disease. Patients will either participate in a three-week cognitive training with concurrent online high-definition tDCS application or placebo ("sham") tDCS or participate in an evidence-based muscle relaxation training combined with placebo tDCS. We hypothesize that cognitive training with sham or active tDCS will result in more pronounced improvement on a transfer task compared to the control group. We also hypothesize that training combined with anodal tDCS will lead to significantly higher performance on a transfer task than training combined with sham tDCS. Additionally, we will determine effects on specifically trained and other untrained cognitive functions immediately after the intervention as well as their maintenance one month later.

ELIGIBILITY:
Inclusion Criteria:

1. History of COVID-19 condition at least 4-6 weeks prior to study inclusion
2. Self-reported concerns regarding cognitive functioning.
3. Age: 18-60 years.

Exclusion Criteria:

1. Acute COVID-19 illness.
2. History of dementia before COVID-19.
3. Other neurodegenerative neurological disorders; epilepsy or history of seizures.
4. Severe and untreated medical conditions that preclude participation in the training, as determined by responsible physician.
5. History of severe alcoholism or use of drugs.
6. Severe psychiatric disorders such as severe depression (if not in remission) or psychosis.
7. Contraindication to tDCS application (Antal et al. 2017).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Working memory performance at post-assessment | 3 weeks
  Percent change of correct responses in the n-back task compared to the pre-training assessment.

SECONDARY OUTCOMES:
Working memory performance at follow-up assessment | 4 weeks after training
  Percent change of correct responses in the n-back task compared to the pre-training assessment.
Working memory training performance (Letter Updating Task) at post-assessment | 3 weeks
  Performance in primary memory training task (Letter Updating Task) at post-assessment, operationalized by number of correctly recalled lists in the letter updating task.
Working memory training performance (Letter Updating Task) at follow-up assessment | 4 weeks after training
  Performance in primary memory training task (Letter Updating Task) at follow-up assessment, operationalized by number of correctly recalled lists in the letter updating task.
Quality of Life at post-assessment | 3 weeks
  PROMIS (Patient-Reported Outcome Measures and Health-Related Quality of Life) score for HRQoL (PROPr score) and scores of subscales (e.g. cognitive function). Every item is rated on scale from 1 to 5, the higher the score the worse the self-reported health evaluation.
Quality of Life at follow-up assessment | 4 weeks after training
  PROMIS (Patient-Reported Outcome Measures and Health-Related Quality of Life) score for HRQoL (PROPr score) and scores of subscales (e.g. cognitive function). Every item is rated on scale from 1 to 5, the higher the score the worse the self-reported health evaluation.
Visuo-spatial performance at post-assessment | 3 weeks
  Visuo-spatial performance at post-assessment operationalized by number of correctly recalled items in the VR task.
Visuo-spatial performance at follow-up assessment | 4 weeks after training
  Visuo-spatial performance at follow-up assessment operationalized by number of correctly recalled items in the VR task.
Post COVID-19 Function at post-assessment | 3 weeks
  Scores of Post COVID-19 Functional Scale (PCFS). PCFS scale grad from 0 (no functional limitations) to 4 (severe functional limitations).
Post COVID-19 Function at follow-up assessment | 4 weeks after training
  Scores of Post COVID-19 Functional Scale (PCFS). PCFS scale grad from 0 (no functional limitations) to 4 (severe functional limitations).

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Prof., Study Director — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be made available to the scientific community upon request.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Thams F, Antonenko D, Fleischmann R, Meinzer M, Grittner U, Schmidt S, Brakemeier EL, Steinmetz A, Floel A. Neuromodulation through brain stimulation-assisted cognitive training in patients with post-COVID-19 cognitive impairment (Neuromod-COV): study protocol for a PROBE phase IIb trial. BMJ Open. 2022 Apr 11;12(4):e055038. doi: 10.1136/bmjopen-2021-055038. PMID 35410927

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-11-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT04944147/SAP_000.pdf